CLINICAL TRIAL: NCT06395389
Title: Development of a Novel Cannabis Brief Intervention for Frequently-Using Emerging Adults: Pilot Randomized Trial
Brief Title: A Brief Intervention for Cannabis Use
Acronym: Bloom
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kathryn Gex, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00133931; K23DA058077 (NIH)
Record Dates: First submitted 2024-04-22; First posted 2024-05-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cannabis Use Disorder
Keywords: Early intervention; Emerging adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Health Education (HealthEdu) (Active Comparator): Brief intervention providing recommendations/advice for good sleep hygiene, nutrition and physical activity, stress, and relationships.
  Interventions: Behavioral: Health Education (HealthEdu)
- Bloom (Experimental): Brief intervention providing personalized discussion of values/goals, reasons for cannabis use, and strategies to help live in line with values and achieve goals.
  Interventions: Behavioral: Bloom

INTERVENTIONS:
Behavioral: Health Education (HealthEdu) — The Health Education condition is a 2-session brief intervention with each session lasting 40-50 minutes and separated by about 1 week (5-10 days). The first session focuses on providing in-depth information on good sleep hygiene and habits to improve sleep and information on positive eating habits, nutrition, and physical activity/functional exercise. The second session focuses on providing information about stress and social connection.
  Other Names: HealthEdu
  Arms: Health Education (HealthEdu)
Behavioral: Bloom — Bloom is a 2-session brief intervention with each session lasting 40-50 minutes and separated by about 1 week (5-10 days). The first session encourages participants to ask themselves what is important to them. This discussion emphasizes identifying values and ways to live in line with their values, as well as why they use cannabis and providing personalized feedback related to their reasons for use. The second session asks participants to reflect on information from session one and consider what they would like to do next to live in line with their values.
  Arms: Bloom

SUMMARY:
The purpose of this study is to compare two brief interventions targeting potentially problematic cannabis use in emerging adults (ages 18-25). Brief interventions are two 40-50 minute sessions separated by 1 week. Eligible emerging adults will complete a detailed cannabis assessment (biological and self-report), followed by one of the two brief interventions, and three follow-up assessments: one immediately after the second session and at 1- and 3-months post-intervention. Assignment to the brief intervention is random. Salivary samples will be collected at baseline, post-intervention, and both follow-ups, for a total of 4 samples, to be tested for tetrahydrocannabinol (THC) and cannabidiol (CBD).

DETAILED DESCRIPTION:
Cannabis is the most widely used federally illicit substance among emerging adults (age 18-25) in the U.S., and frequent cannabis use is associated with myriad long-term health, social, and academic/occupational consequences. Despite this, rates of perceived risk of daily/regular cannabis use have steadily declined over the past two decades, and this is associated with increased frequency of use, a risk for for Cannabis Use Disorder (CUD). Brief interventions (BIs) are among the most frequently used approaches for addressing problematic or potentially problematic substance use in non-treatment-seeking adolescents and young adults. Although several cannabis brief interventions have been developed and tested to date, meta-analyses indicate that the efficacy of these interventions for emerging adults is mixed and the quality of studies is low, suggesting that novel approaches and rigorous methodology are necessary to improve efficacy. The current study will evaluate the feasibility, acceptability, and preliminary efficacy of a novel cannabis BI for emerging adults who frequently use cannabis.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-25
* Self-Report report cannabis use on at least 20 days of the past 30 days.
* Completion of an Intake Visit (PRO #94743)
* Submit a positive urine cannabinoid test during the Intake Visit

Exclusion Criteria:

* Currently engaged in substance use treatment for any type of substance use or currently treatment seeking
* History of substance use treatment for any type of substance
* Severe alcohol use disorder or presence of any substance use disorder (SUD) requiring a higher level of care
* Significant or acutely unstable medical or psychiatric problems (i.e., psychosis, mania) that would contraindicate research procedures, interfere with safety, compromise data integrity, or preclude consistent study participation
* Significant risk of suicide or homicide

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Timeline Followback (TLFB) | Baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  The TLFB is a calendar based assessment that is able to capture the frequency and quantity of substance use and other measurable behaviors. Responders identify anchor dates to facilitate recall of days in which substances were used.

SECONDARY OUTCOMES:
Marijuana Assessment of Problems Inventory (MAPI) | Baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  This is a 23-item assessment of the frequency in which problems or negative consequences associated with cannabis use have occurred. For each item, participants select 0 times, 1-2 times, 3-5 times, 6-10 times, or 10+ times in the past month. Higher scores on this inventory indicate a higher frequency of problems or consequences experienced.
Mini International Neuropsychiatric Interview (MINI) Cannabis Use Disorder Module | Baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  This is a 12-item semi-structured clinician interview that assesses diagnostic symptom criteria of cannabis use disorder (CUD) from the Diagnostic and Statistical Manual 5th Edition (DSM-5). Clinicians select either 'yes' or 'no' for the presence of the symptom.
Oral Fluid Biospecimen Assay | Baseline, 2-week follow-up, 1-month follow-up, 3-month follow-up, 6-month follow-up
  This is a relatively brief objective assessment of recent cannabis use that is collected through mouth swab and is tested at Forensic Fluids Laboratory for the presence of delta-9 tetrahydrocannabinol (THC), delta-8 THC, and cannabidiol (CBD) using a cut-off of 1 nanogram/liter.

OTHER OUTCOMES:
Comprehensive Marijuana Motives Questionnaire (CMMQ) | Baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  This is a 44-item measure capturing the various reasons why the individual uses cannabis, including for enjoyment/enhancement, coping, social anxiety, sleep, celebration, boredom, conformity, expansion, and others. For each item, participants select 1 (almost never/never), 2 (some of the time), 3 (half the time), 4 (most of the time), or 5 (almost always/always). Higher average scores indicate more reasons for cannabis use / using cannabis more often for identified reasons.
Protective Behavioral Strategies - Marijuana (PBSM) | Baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  This is a 36-item measure that assesses the use of different cognitive and behavioral strategies that are intended to minimize harms or negative consequences associated with cannabis use. For each item, participants select 1 (Never), 2 (Rarely), 3 (Occasionally), 4 (Sometimes), 5 (Usually), or 6 (Always). Higher scores indicate more frequent use of strategies to reduce the risk of harm or negative consequences from cannabis use.
Consideration of Future Consequences Scale (CFCS) | Baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  This is a 12-item scale that assesses how characteristic or uncharacteristic it is for the individual to take into account the future consequences of an action or choice made in the present moment. Participants rate each item from 1 to 5: 1 (extremely uncharacteristic), 2 (somewhat uncharacteristic), 3 (uncertain), 4 (somewhat characteristic), 5 (extremely characteristic). Higher scores indicate a greater consideration of future consequences.
The Adolescent Reinforcement Survey Schedule - Substance Use Version (ARSS-SUV) | Baseline, 1-month follow-up, 3-month follow-up, 6-month follow-up
  This is a 35-item assessment of day-to-day activities that individuals engage in with or without the use of substances (in this case cannabis) and the extent to which they enjoyed participating in the activity with or without substance use. For each frequency item, participants select 0 (not engaged), 1 (once a week or less), 2 (2-4 times per week), 3 (about once a day), or 4 (more than once a day). For each enjoyment item, participants select (0 (unpleasant/neutral), 1 (mildly pleasant), 2 (moderately pleasant), 3 (very pleasant), or 4 (extremely pleasant). A cross-product of frequency and enjoyment is created for each item to calculate final scores of substance-free reinforcement and substance-related reinforcement. A reinforcement ratio is then calculated for substance-free and substance-related activities by dividing each score from the sum of both scores (i.e., substance-free / (substance-free + substance-related); or substance-related / (substance-free + substance-related)).

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Gex, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No